CLINICAL TRIAL: NCT01113944
Title: Training in the Workplace
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Sara W Lazar, Associate Research Scientist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: YEL1
Record Dates: First submitted 2010-04-28; First posted 2010-04-30 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: Healthy Individuals

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Program 1 (Active Comparator): Program 1
  Interventions: Behavioral: Program 1
- Program 2 (Active Comparator): Program 2
  Interventions: Behavioral: Program 2

INTERVENTIONS:
Behavioral: Program 1
  Arms: Program 1
Behavioral: Program 2
  Arms: Program 2

SUMMARY:
We are testing whether various cognitive training procedures can enhance cognition and brain function

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals aged 18-50 years old
* Right handed
* Must have reliable internet access from a desktop computer with webcam
* English speaking

Exclusion Criteria:

* Neurological conditions
* pregnancy
* metalic implants

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2010-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
MRI | 2 hours Pre and Post intervention
  Functional and structural MR images will be acquired

CONTACTS AND LOCATIONS:
Overall Officials: Sara Lazar, PhD, Principal Investigator — MGH
Locations (1):
- Massachusettts General Hospital, Boston, Massachusetts, United States